CLINICAL TRIAL: NCT03574662
Title: A Prospective Trial to Evaluate the Utility of Focused Frailty Interventions on Patients With Advanced Heart Failure
Brief Title: The Utility of Focused Frailty Interventions on Patients With Advanced Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sudhir Kushwaha, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-000665
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: frailty; advanced
MeSH Terms: conditions — Heart Failure; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frailty assessment in Advanced heart failure (Experimental): Subjects with advanced heart failure defined as current or recent (within the last 3 months) New York Heart Association (NYHA) class III or IV symptoms.
  Interventions: Other: Frailty assessment; Other: Quality of life assessment

INTERVENTIONS:
Other: Frailty assessment — This assessment consists of a combination of gait speed measurement via infrared sensors as well as a grip strength assessment. Patients will then attend cardiac rehabilitation for an abbreviated six week program.
Other: Quality of life assessment — This assessment consists of two questionnaires, Kansas City Cardiomyopathy Questionnaire and Minnesota Living with Heart Failure questionnaire. Patients will then attend cardiac rehabilitation for an abbreviated six week program.

SUMMARY:
The Researchers are doing this study to find out if the cardiac rehabilitation program can improve measurements of frailty and improve independence, functional abilities, and feelings about health. Frailty can be measured by weakness (as measured by hand grip strength), slowness (as measured by walking speed), low level of physical activity, low energy or self-reported exhaustion, and unintentional weight loss.

DETAILED DESCRIPTION:
Participants with advanced heart failure with a New York Heart Association class of III or IV symptoms within the last 3 months will be identified by either their outpatient heart failure clinic notes or inpatient cardiology notes. Patients will be approached for participation if cardiac rehab is mentioned in the notes and inclusion/exclusion criteria it met. Once the consent is signed, the baseline visit will be scheduled, this will be done before cardiac rehab has started. The baseline visit include frailty assessment measured by a walk time/gait speed test and handgrip strength test, and quality of life assessment measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) and Minnesota Living with Heart Failure (MLHF) questionnaire. Patients will then attend cardiac rehabilitation for six week program. The cardiac rehab program will be designed by the individual facility due to the variation in exercise tolerance of each patient, no universal protocol will be used. After the six weeks of cardiac rehab, up to 16 weeks post-completion, the patient will return to Mayo Clinic Rochester to complete the frailty and quality of life assessment.

ELIGIBILITY:
Inclusion criteria:

* Advanced heart failure patients.
* These include patients with Current NYHA class III-IV symptoms at the current time or within the preceding three months.
* Outpatient heart failure clinic with mention of cardiac rehab in patient medical record in the past year OR patients admitted to the hospital to any inpatient cardiology service (including the coronary care unit (CCU)) and mention of cardiac rehab from service.

Exclusion criteria:

* Unable to perform physical activities due to anatomic or musculoskeletal comorbidities
* Physical activity is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in gait speed | baseline, 6 weeks
  The time it takes to walk a specified distance, as measured in meters per second
Change in hand grip | baseline, 6 weeks
  The amount of force that the hand can squeeze, as measured in kilograms
Change in Kansas City Cardiomyopathy Questionnaire | baseline, 6 weeks
  The KCCQ is a 23-item questionnaire that quantifies dyspnea, fatigue, and edema on physical, social, and emotional functions of the patient. Responses are categorized by 3 subscales (burden, limitations, and quality of life) with a possible range of scores from 0 to 100, 100 being the least burdened by their symptoms. This questionnaire independently measures the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social functions, and how their heart failure impacts their quality of life within a two week recall period.
Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) | baseline, 6 weeks
  The MLHFQ asks each person to indicate using a 6-point (zero to five) Likert scale how much each of 21 facets prevents them from living as they desire. The questionnaire assesses the impact of frequent physical symptoms - shortness of breath, fatigue, peripheral edema, and difficulty sleeping - and psychological symptoms of anxiety and depression. In addition, the effects of heart failure on physical and social functioning are incorporated into the measure. Since treatments might have side effects in addition to ameliorating symptoms and functional limitations produced by heart failure, questions about side effects of medications, hospital stays and costs of care are also included to help measure the overall impact of a treatment on quality of life. Although the MLHFQ incorporates relevant aspects of the key dimensions of quality of life, the questionnaire was not designed to measure any particular dimension separately.

SECONDARY OUTCOMES:
Delay in Left Ventricular Assist Device (LVAD) placement | 16 weeks
  Number of days until LVAD placement
Post surgical length of stay | 16 weeks
  Number of days subject in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir S Kushwaha, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh M, Stewart R, White H. Importance of frailty in patients with cardiovascular disease. Eur Heart J. 2014 Jul;35(26):1726-31. doi: 10.1093/eurheartj/ehu197. Epub 2014 May 26. PMID 24864078
- [Background] Kulminski AM, Ukraintseva SV, Culminskaya IV, Arbeev KG, Land KC, Akushevich L, Yashin AI. Cumulative deficits and physiological indices as predictors of mortality and long life. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1053-9. doi: 10.1093/gerona/63.10.1053. PMID 18948555
- [Background] Kulminski AM, Ukraintseva SV, Kulminskaya IV, Arbeev KG, Land K, Yashin AI. Cumulative deficits better characterize susceptibility to death in elderly people than phenotypic frailty: lessons from the Cardiovascular Health Study. J Am Geriatr Soc. 2008 May;56(5):898-903. doi: 10.1111/j.1532-5415.2008.01656.x. Epub 2008 Mar 21. PMID 18363679
- [Background] Dunlay SM, Park SJ, Joyce LD, Daly RC, Stulak JM, McNallan SM, Roger VL, Kushwaha SS. Frailty and outcomes after implantation of left ventricular assist device as destination therapy. J Heart Lung Transplant. 2014 Apr;33(4):359-65. doi: 10.1016/j.healun.2013.12.014. Epub 2013 Dec 27. PMID 24486165
- [Background] Amrock LG, Deiner S. The implication of frailty on preoperative risk assessment. Curr Opin Anaesthesiol. 2014 Jun;27(3):330-5. doi: 10.1097/ACO.0000000000000065. PMID 24566452
- [Background] Thalji NM, Suri RM, Greason KL, Schaff HV. Risk assessment methods for cardiac surgery and intervention. Nat Rev Cardiol. 2014 Dec;11(12):704-14. doi: 10.1038/nrcardio.2014.136. Epub 2014 Sep 23. PMID 25245832
- [Background] Flint KM, Matlock DD, Lindenfeld J, Allen LA. Frailty and the selection of patients for destination therapy left ventricular assist device. Circ Heart Fail. 2012 Mar 1;5(2):286-93. doi: 10.1161/CIRCHEARTFAILURE.111.963215. No abstract available. PMID 22438521
- [Background] Rockwood K, Andrew M, Mitnitski A. A comparison of two approaches to measuring frailty in elderly people. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):738-43. doi: 10.1093/gerona/62.7.738. PMID 17634321
- [Background] Chung CJ, Wu C, Jones M, Kato TS, Dam TT, Givens RC, Templeton DL, Maurer MS, Naka Y, Takayama H, Mancini DM, Schulze PC. Reduced handgrip strength as a marker of frailty predicts clinical outcomes in patients with heart failure undergoing ventricular assist device placement. J Card Fail. 2014 May;20(5):310-5. doi: 10.1016/j.cardfail.2014.02.008. Epub 2014 Feb 22. PMID 24569037
- [Background] Flint KM, Matlock DD, Sundareswaran KS, Lindenfeld J, Spertus JA, Farrar DJ, Allen LA. Pre-operative health status and outcomes after continuous-flow left ventricular assist device implantation. J Heart Lung Transplant. 2013 Dec;32(12):1249-54. doi: 10.1016/j.healun.2013.09.005. Epub 2013 Oct 8. PMID 24119729
- [Background] Binder EF, Schechtman KB, Ehsani AA, Steger-May K, Brown M, Sinacore DR, Yarasheski KE, Holloszy JO. Effects of exercise training on frailty in community-dwelling older adults: results of a randomized, controlled trial. J Am Geriatr Soc. 2002 Dec;50(12):1921-8. doi: 10.1046/j.1532-5415.2002.50601.x. PMID 12473001
- [Background] Cesari M, Vellas B, Hsu FC, Newman AB, Doss H, King AC, Manini TM, Church T, Gill TM, Miller ME, Pahor M; LIFE Study Group. A physical activity intervention to treat the frailty syndrome in older persons-results from the LIFE-P study. J Gerontol A Biol Sci Med Sci. 2015 Feb;70(2):216-22. doi: 10.1093/gerona/glu099. Epub 2014 Nov 11. PMID 25387728
- [Background] Clegg A, Barber S, Young J, Iliffe S, Forster A. The Home-based Older People's Exercise (HOPE) trial: a pilot randomised controlled trial of a home-based exercise intervention for older people with frailty. Age Ageing. 2014 Sep;43(5):687-95. doi: 10.1093/ageing/afu033. Epub 2014 Apr 16. PMID 24742587
- [Background] Molino-Lova R, Pasquini G, Vannetti F, Paperini A, Forconi T, Polcaro P, Zipoli R, Cecchi F, Macchi C. Effects of a structured physical activity intervention on measures of physical performance in frail elderly patients after cardiac rehabilitation: a pilot study with 1-year follow-up. Intern Emerg Med. 2013 Oct;8(7):581-9. doi: 10.1007/s11739-011-0654-z. Epub 2011 Jul 9. PMID 21744061
- [Background] Peterson MJ, Sloane R, Cohen HJ, Crowley GM, Pieper CF, Morey MC. Effect of telephone exercise counseling on frailty in older veterans: project LIFE. Am J Mens Health. 2007 Dec;1(4):326-34. doi: 10.1177/1557988307306153. Epub 2007 Oct 3. PMID 19482814
- [Background] Chan DC, Tsou HH, Yang RS, Tsauo JY, Chen CY, Hsiung CA, Kuo KN. A pilot randomized controlled trial to improve geriatric frailty. BMC Geriatr. 2012 Sep 25;12:58. doi: 10.1186/1471-2318-12-58. PMID 23009149
- [Background] Villareal DT, Banks M, Sinacore DR, Siener C, Klein S. Effect of weight loss and exercise on frailty in obese older adults. Arch Intern Med. 2006 Apr 24;166(8):860-6. doi: 10.1001/archinte.166.8.860. PMID 16636211
- [Background] Fragala MS, Dam TT, Barber V, Judge JO, Studenski SA, Cawthon PM, McLean RR, Harris TB, Ferrucci L, Guralnik JM, Kiel DP, Kritchevsky SB, Shardell MD, Vassileva MT, Kenny AM. Strength and function response to clinical interventions of older women categorized by weakness and low lean mass using classifications from the Foundation for the National Institute of Health sarcopenia project. J Gerontol A Biol Sci Med Sci. 2015 Feb;70(2):202-9. doi: 10.1093/gerona/glu110. Epub 2014 Aug 18. PMID 25135999
- [Background] Marsh AP, Chmelo EA, Katula JA, Mihalko SL, Rejeski WJ. Should physical activity programs be tailored when older adults have compromised function? J Aging Phys Act. 2009 Jul;17(3):294-306. doi: 10.1123/japa.17.3.294. PMID 19799101